CLINICAL TRIAL: NCT07247955
Title: Effectiveness of the Guided and Traditional Cognitive Behavioral Therapy Protocol in a Patient With Treatment-resistant Panic Disorder
Brief Title: Guided and Traditional Cognitive Behavioral Therapy Protocol for Resistant Panic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Luisa Pelucio Ribeiro Barbosa, Master - Principal Investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: UFRJ-2025-001
Record Dates: First submitted 2025-05-22; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-05

CONDITIONS: Panic Disorder
Keywords: Panic disorder; Cognitive behavioral therapy; Application
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Intervention Model Description: As a pilot study comparing two groups of patients with PD in different forms of care, the data from 23 patients with panic disorder undergoing traditional CBT and 23 patients with panic disorder doing self-guided therapy through an application were collected. The groups were randomized, they had no comorbidities, all patients were undergoing psychiatric follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of 23 patients undergoing traditional cognitive behavioral therapy (Experimental): Twenty-three patients were selected for group. The group consisted of patients with panic disorder and breathing difficulties in a traditional cognitive behavioral therapy format, 8-session treatment protocol.
  Interventions: Behavioral: The group intervention used the sessions described in traditional form
- Group of 23 patients undergoing self-guided cognitive behavioral therapy using an app (Experimental): Twenty-three patients were selected for group. The group consisted of patients with panic disorder and breathing difficulties in a self-guided cognitive behavioral therapy format, using the 8-session treatment protocol.
  Interventions: Behavioral: The group intervention used the sessions described in a self-guided format using an application

INTERVENTIONS:
Behavioral: The group intervention used the sessions described in traditional form — Model of the sessions:
  * Session 1 - General information for the Client
  * Session 2 - Breaking the panic cycle
  * Session 3 - Increasing the range of cognitive management skills
  * Session 4 - Improving corporal management skills
  * Session 5 - Strengthening self-efficacy
  * Session 6 - Stimulating life reorientation
  * Session 7 - Promoting existential management
  * Session 8 - Revising and evaluating the treatment
  Arms: Group of 23 patients undergoing traditional cognitive behavioral therapy
Behavioral: The group intervention used the sessions described in a self-guided format using an application — Model of the sessions:
  * Session 1 - General information for the Client
  * Session 2 - Breaking the panic cycle
  * Session 3 - Increasing the range of cognitive management skills
  * Session 4 - Improving corporal management skills
  * Session 5 - Strengthening self-efficacy
  * Session 6 - Stimulating life reorientation
  * Session 7 - Promoting existential management
  * Session 8 - Revising and evaluating the treatment
  Arms: Group of 23 patients undergoing self-guided cognitive behavioral therapy using an app

SUMMARY:
Self-guided therapy for anxiety disorders has focused on various cognitive-behavioral treatments mediated by technologies such as web applications. This study aims to compare two groups of patients with panic disorder undergoing two clinical psychological treatment models: one traditional cognitive behavioral therapy (CBT), and the other self-guided CBT using a digital application.

An application was developed in which both treatment models follow the same eight-session CBT manual. Patients are evaluated using psychological assessments at the first and eighth sessions.

The study includes 46 patients divided into two groups of 23 participants each. Both groups undergo individual assessments at the beginning and end of the treatment protocol.

DETAILED DESCRIPTION:
As such, an application was developed whereby the two models follow the same treatment manual of eight sessions, with the patients being evaluated using psychological tests at the first and eighth sessions.

Methods: A total of 46 patients were separated into two groups of 23 patients, one in each format, with the patients in both groups being individually evaluated at their first and eighth sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IPUB screening through the panic and respiratory laboratory outpatient clinic.
* Diagnosis of panic disorder confirmed.
* Age between 18 and 60 years.
* Under psychiatric follow-up by a university psychiatrist and taking medication.
* Provide written informed consent to participate and have data stored.

Exclusion Criteria:

* Patients without a diagnosis of panic disorder.
* Age under 18 or over 60 years.
* Not undergoing psychiatric follow-up.
* Presence of other psychiatric or medical diagnoses.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Efficacy criteria | Baseline (Week 1) and Post-intervention (Week 8)
  Primary Outcome Measure 1 Title: Beck Anxiety Inventory (BAI) total score Time Frame: Baseline (Week 1) and Post-intervention (Week 8) Description: The BAI is a 21-item self-report questionnaire that measures the severity of anxiety symptoms. Total scores range from 0 to 63; higher scores indicate greater anxiety. Administered to all participants in both groups. Results will be reported separately for each time point.
  Unit of Measure: Points on a scale (0-63) Primary Outcome Measure 2 Title: Beck Depression Inventory (BDI) total score Time Frame: Baseline (Week 1) and Post-intervention (Week 8) Description: The BDI is a 21-item self-report inventory assessing depressive symptoms. Scores range from 0 to 63, with higher scores indicating greater severity of depression. Applied to all participants in both groups, with separate reporting for each assessment.
  Unit of Measure: Points on a scale (0-63)

SECONDARY OUTCOMES:
Efficacy criteria | Baseline (Week 1) and Post-intervention (Week 8)
  Outcome Measure 3 Title: Mindful Attention Awareness Scale (MAAS) total score Time Frame: Baseline (Week 1) and Post-intervention (Week 8) Description: The MAAS is a 15-item scale measuring mindfulness in daily life. Scores range from 15 to 90; higher scores reflect greater mindfulness. Administered to all participants. Scores will be reported separately at each time point.
  Unit of Measure: Points on a scale (15-90) Outcome Measure 4 Title: Brief Resilient Coping Scale (BRCS) total score Time Frame: Baseline (Week 1) and Post-intervention (Week 8) Description: The BRCS is a 4-item scale assessing the tendency to cope with stress in a resilient manner. Scores range from 4 to 20; higher scores indicate more adaptive coping. Administered to both groups. Each time point reported separately.
  Unit of Measure: Points on a scale (4-20)

OTHER OUTCOMES:
Efficacy criteria | Baseline (Week 1) and Post-intervention (Week 8)
  Outcome Measure 5 Title: WHOQOL-BREF domain scores - Physical, Social, Environmental Time Frame: Baseline (Week 1) and Post-intervention (Week 8) Description: The WHOQOL-BREF assesses quality of life. This outcome includes scores from the Physical Health, Social Relationships, and Environment domains. Each domain score ranges from 4 to 20; higher scores represent better quality of life.
  Unit of Measure: Points on a scale (4-20) Outcome Measure 6 Title: Panic and Agoraphobia Scale (PAS) total score Time Frame: Baseline (Week 1) and Post-intervention (Week 8) Description: The PAS is a clinician-administered scale with 13 items assessing the severity of panic and agoraphobia symptoms. Scores range from 0 to 52; higher scores indicate more severe symptoms. Applied to all participants.
  Unit of Measure: Points on a scale (0-52)

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Pelucio, Master, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Universidade Federal do Rio de JAneiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gal E, Stefan S, Cristea IA. The efficacy of mindfulness meditation apps in enhancing users' well-being and mental health related outcomes: a meta-analysis of randomized controlled trials. J Affect Disord. 2021 Jan 15;279:131-142. doi: 10.1016/j.jad.2020.09.134. Epub 2020 Oct 7. PMID 33049431
- [Result] Yogeswaran V, El Morr C. Effectiveness of online mindfulness interventions on medical students' mental health: a systematic review. BMC Public Health. 2021 Dec 18;21(1):2293. doi: 10.1186/s12889-021-12341-z. PMID 34920715
- [Result] Linardon J. Can Acceptance, Mindfulness, and Self-Compassion Be Learned by Smartphone Apps? A Systematic and Meta-Analytic Review of Randomized Controlled Trials. Behav Ther. 2020 Jul;51(4):646-658. doi: 10.1016/j.beth.2019.10.002. Epub 2019 Nov 26. PMID 32586436
- [Result] Whittaker R, McRobbie H, Bullen C, Borland R, Rodgers A, Gu Y. Mobile phone-based interventions for smoking cessation. Cochrane Database Syst Rev. 2012 Nov 14;11:CD006611. doi: 10.1002/14651858.CD006611.pub3. PMID 23152238
- [Result] Bakker D, Kazantzis N, Rickwood D, Rickard N. Mental Health Smartphone Apps: Review and Evidence-Based Recommendations for Future Developments. JMIR Ment Health. 2016 Mar 1;3(1):e7. doi: 10.2196/mental.4984. PMID 26932350
- [Result] Loucas CE, Fairburn CG, Whittington C, Pennant ME, Stockton S, Kendall T. E-therapy in the treatment and prevention of eating disorders: A systematic review and meta-analysis. Behav Res Ther. 2014 Dec;63:122-31. doi: 10.1016/j.brat.2014.09.011. Epub 2014 Oct 5. PMID 25461787
- [Result] Schueller SM, Torous J. Scaling evidence-based treatments through digital mental health. Am Psychol. 2020 Nov;75(8):1093-1104. doi: 10.1037/amp0000654. PMID 33252947
- [Result] Wu J, Ma Y, Zuo Y, Zheng K, Zhou Z, Qin Y, Ren Z. Effects of Mindfulness Exercise Guided by a Smartphone App on Negative Emotions and Stress in Non-Clinical Populations: A Systematic Review and Meta-Analysis. Front Public Health. 2022 Jan 25;9:773296. doi: 10.3389/fpubh.2021.773296. eCollection 2021. PMID 35155341
- [Result] Rathbone AL, Clarry L, Prescott J. Assessing the Efficacy of Mobile Health Apps Using the Basic Principles of Cognitive Behavioral Therapy: Systematic Review. J Med Internet Res. 2017 Nov 28;19(11):e399. doi: 10.2196/jmir.8598. PMID 29187342
- [Result] Hansen WB, Scheier LM. Specialized Smartphone Intervention Apps: Review of 2014 to 2018 NIH Funded Grants. JMIR Mhealth Uhealth. 2019 Jul 29;7(7):e14655. doi: 10.2196/14655. PMID 31359866
- [Result] Hwang WJ, Ha JS, Kim MJ. Research Trends on Mobile Mental Health Application for General Population: A Scoping Review. Int J Environ Res Public Health. 2021 Mar 2;18(5):2459. doi: 10.3390/ijerph18052459. PMID 33801537
- [Result] Firth J, Torous J, Carney R, Newby J, Cosco TD, Christensen H, Sarris J. Digital Technologies in the Treatment of Anxiety: Recent Innovations and Future Directions. Curr Psychiatry Rep. 2018 May 19;20(6):44. doi: 10.1007/s11920-018-0910-2. PMID 29779065
- [Result] Wright JH, Mishkind M, Eells TD, Chan SR. Computer-Assisted Cognitive-Behavior Therapy and Mobile Apps for Depression and Anxiety. Curr Psychiatry Rep. 2019 Jun 27;21(7):62. doi: 10.1007/s11920-019-1031-2. PMID 31250242
- [Result] Khademian F, Aslani A, Bastani P. The effects of mobile apps on stress, anxiety, and depression: overview of systematic reviews. Int J Technol Assess Health Care. 2020 Dec 14;37:e4. doi: 10.1017/S0266462320002093. PMID 33314997
- [Result] Ito LM, Noshirvani H, Basoglu M, Marks IM. Does exposure to internal cues enhance exposure to external cues in agoraphobia with panic? A pilot controlled study of self-exposure. Psychother Psychosom. 1996;65(1):24-28. doi: 10.1159/000289027. PMID 8838693
- [Result] Ito LM, de Araujo LA, Tess VL, de Barros-Neto TP, Asbahr FR, Marks I. Self-exposure therapy for panic disorder with agoraphobia: randomised controlled study of external v. interoceptive self-exposure. Br J Psychiatry. 2001 Apr;178:331-6. doi: 10.1192/bjp.178.4.331. PMID 11282812
- [Result] Clark DM. A cognitive approach to panic. Behav Res Ther. 1986;24(4):461-70. doi: 10.1016/0005-7967(86)90011-2. No abstract available. PMID 3741311